CLINICAL TRIAL: NCT01099696
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Evaluate the Benefit of a Probiotic (Bifidobacterium Infantis 35624) in Healthy Subjects With a History of Abdominal Discomfort and Bloating
Brief Title: Study to Evaluate a Probiotic in Healthy Subjects With a History of Abdominal Discomfort and Bloating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009120
Record Dates: First submitted 2010-04-06; First posted 2010-04-07 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Abdominal Discomfort; Bloating
Keywords: abdominal discomfort and bloating

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- B. infantis 35624 (Experimental): B. infantis 35624 in white capsules
  Interventions: Dietary Supplement: B. infantis 35624
- placebo (Placebo Comparator): white placebo capsules (inert)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: B. infantis 35624 — B. infantis 35624 in white capsules
  Arms: B. infantis 35624
Dietary Supplement: placebo — white placebo capsules
  Arms: placebo

SUMMARY:
This is a multicenter, double-blind, randomized, placebo-controlled, 6-week study of a probiotic for abdominal discomfort and bloating in healthy subjects.

DETAILED DESCRIPTION:
This is a multicenter, double-blind, randomized, placebo-controlled, parallel-group, 6-week study of a probiotic for abdominal discomfort and bloating in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* healthy men and non-pregnant, non-lactating women aged 18 to 75 years of age;
* Body Mass Index (BMI) < or = 40;
* if female, postmenopausal or using adequate contraception
* if over 50 years of age, have had a colonoscopy performed in the previous 5 years with findings that are normal for this population
* be willing to refrain from taking dietary supplements or other foods that contain fermented live bacteria during the study and be willing to refrain from taking any medications or preparations that treat lower digestive upsets
* have experienced abdominal discomfort and bloating at least twice a week, on average, over the last 3 months.

Exclusion Criteria:

* have been under a physician's care for functional bowel disorders within the past year or have taken prescription medication for functional bowel disorders within the past year;
* have alarm symptoms suggestive of an underlying disease;
* have prior GI surgery (appendectomy and hernia repair are not excluded and cholecystectomy at least 3 years ago is not excluded);
* have a significant acute or chronic coexisting illness or condition;
* have used systemic steroidal agents within the last 30 days;
* have used oral or systemic antibiotics within the last 30 days;
* have used probiotics at least 3 times a week within the last 30 days;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2010-04; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The change in abdominal discomfort and bloating | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jose Brum, MD, Study Director — P&G
Locations (10):
- United States (10):
  - Research Site, Chicago, Illinois
  - Research Site, Rockford, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Chevy Chase, Maryland
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Greer, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Charlottesville, Virginia

REFERENCES:
- [Derived] Ringel-Kulka T, McRorie J, Ringel Y. Multi-Center, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study to Evaluate the Benefit of the Probiotic Bifidobacterium infantis 35624 in Non-Patients With Symptoms of Abdominal Discomfort and Bloating. Am J Gastroenterol. 2017 Jan;112(1):145-151. doi: 10.1038/ajg.2016.511. Epub 2016 Nov 15. PMID 27845337